CLINICAL TRIAL: NCT03019757
Title: Distinguishing Between Alzheimer's Disease, Lewy Body Dementia, and Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Douglas Scharre (Other)
Collaborators: Avid Radiopharmaceuticals (Industry); Mangurian Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Douglas Scharre, Professor, Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2014H0415
Record Dates: First submitted 2015-09-03; First posted 2017-01-13 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease; Lewy Body Dementia; Parkinson's Disease
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Parkinson Disease | interventions — ioflupane; florbetapir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants will have the option to participate in a lumbar puncture sub-study as well as a brain donation program. These samples will be retained in the Buckeye Biospecimen Repository or the Buckeye Brain Bank, respectively.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alzheimer's disease: Individuals with a clinical diagnosis of Alzheimer's disease will undergo the interventions including DaTscan, F18-AV-45, FDG-PET, APOE genotype, Polysomnogram, and Clinical Assessment.
  Interventions: Radiation: DaTscan; Radiation: F18-AV-45; Radiation: FDG-PET; Genetic: APOE genotype; Procedure: Polysomnogram; Behavioral: Clinical Assessment
- Lewy Body dementia: Individuals with a clinical diagnosis of Lewy Body Dementia will undergo the interventions including DaTscan, F18-AV-45, FDG-PET, APOE genotype, Polysomnogram, and Clinical Assessment.
  Interventions: Radiation: DaTscan; Radiation: F18-AV-45; Radiation: FDG-PET; Genetic: APOE genotype; Procedure: Polysomnogram; Behavioral: Clinical Assessment
- Parkinson's disease: Individuals with a clinical diagnosis of Parkinson's disease will undergo the interventions including DaTscan, F18-AV-45, FDG-PET, APOE genotype, Polysomnogram, and Clinical Assessment.
  Interventions: Radiation: DaTscan; Radiation: F18-AV-45; Radiation: FDG-PET; Genetic: APOE genotype; Procedure: Polysomnogram; Behavioral: Clinical Assessment

INTERVENTIONS:
Radiation: DaTscan — A functional imaging of the dopamine transporter using the radioligand [123I]FP-CIT
Radiation: F18-AV-45 — A brain scan to to measure the extent of amyloid deposition
Radiation: FDG-PET — a brain scan measuring total and regional cerebral glucose metabolism wtih positron emission tomographs with 2-(18F)
Genetic: APOE genotype — 10 ml of whole blood will be drawn and shipped to Athena Diagnostics for genetic testing.
Procedure: Polysomnogram — Overnight sleep study
Behavioral: Clinical Assessment — Clinical assessments include cognitive, behavioral, and motor evaluations

SUMMARY:
The study is designed to characterize the clinical, neuropsychological, polysomnographic, and neuroimaging findings among subjects with Alzheimer's disease, Lewy Body dementia, and Parkinsons' Disease.

DETAILED DESCRIPTION:
The study will use structural and functional MRIs, daTscans, fluorodeoxyglucose (FDG) PET scans, Amyvid PET scans, polysomnographs, neuropsychological testing, cerebrospinal fluid in willing participants to distinguish between a diagnosis of Alzheimer's disease, Lewy Body dementia, and Parkinson's Disease. All subjects will have a clinical evaluation, physical examination including vital signs and orthostatic blood pressures and pulses, neurological examination including UPDRS evaluation, genetic blood sample collection, neuropsychological testing, polysomnogram, and neuroimaging. The study partner will also be interviewed for completion of all of the behavioral and functional measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the standard clinical criteria of the syndromes of interest
* All subjects must have enough cognitive abilities to complete study procedures, which will be operationally defined as having a Mini Mental State Examination (MMSE) score greater or equal to 10.
* Subjects must be on stable cognitive and psychoactive medication regimen for the preceding four weeks of enrollment.
* Subjects must have a responsible study partner that either lives with them or is in regular contact with them at least 4 out of 7 days per week.
* Subjects must have visual and auditory acuity adequate for testing.

Exclusion Criteria:

* Any other condition (other than the primary diagnosis), which in the opinion of the investigators might contribute to the syndrome of dementia or complicate its assessment.
* active medical disorder that could preclude participation in this protocol
* Women who are pregnant or are breast feeding
* severe renal impairment as defined by glomerular filtration rate (GFR) less than 30 (may have increased radiation exposure with the DaTscan).
* Subjects in whom English is not the 1st language
* Subjects with educational level less than 12 years
* Subjects who have ever participated in an experimental study with an amyloid targeting agent unless it can be documented that the subject received only placebo during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must have a clinical diagnosis of either Alzheimer's disease, Lewy Body Dementia, or Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE-1) | Baseline
  Global neuropsychological measure
Wechsler Adult Intelligence Scale 4th edition (WAIS-4) Vocabulary | Baseline
  Neuropsychological measure of premorbid IQ estimate
Wechsler Adult Intelligence Scale 4th edition (WAIS-4) Digit Span | Baseline
  Neuropsychological measure of attention
Wechsler Adult Intelligence Scale 4th edition (WAIS-4) Block Design | Baseline
  Neuropsychological measure of visuospatial perception/ reasoning
Wechsler Adult Intelligence Scale 4th edition (WAIS-4) Matrix Reasoning | Baseline
  Neuropsychological measure of executive functioning
Wechsler Adult Intelligence Scale 4th edition (WAIS-4) Reliable Digits (embedded measure) | Baseline
  Neuropsychological measure of effort
Wechsler Memory Scale 3rd ed. (WAIS-3) Spatial Span | Baseline
  Neuropsychological measure of attention
Wechsler Memory Scale 3rd ed. (WAIS-3) Logical Memory 1 & 2 | Baseline
  Neuropsychological measure of memory
Trail Making Test A | Baseline
  Neuropsychological measure of executive functioning/psychomotor processing speed
Trail Making Test B | Baseline
  Neuropsychological measure of executive functioning
Boston Naming Test | Baseline
  Neuropsychological measure of language
Controlled Oral Word Association Test (COWAT)- Animal Naming | Baseline
  Neuropsychological measure of language/verbal fluency
Judgment of Line Orientation Standardized Test | Baseline
  Neuropsychological measure of visuospatial perception/ reasoning
Brief Visuospatial Memory Test (BVMT) | Baseline
  Neuropsychological measure of memory
California Verbal Learning Test (CVLT-2) | Baseline
  Neuropsychological measure of memory
Wisconsin Card Sorting Task | Baseline
  Neuropsychological measure of executive functioning
California Verbal Learning Test (CVLT-2) Forced Choice (embedded measure) | Baseline
  Neuropsychological measure of effort
Self Administered Gerocognitive Examination- A brief cognitive assessment instrument for mild cognitive impairment and early dementia | Baseline
  Global neuropsychological measure
Apolipoprotein E (APOE) Genotyping of a whole blood sample | Baseline
  10 ml of whole blood will be drawn for APOE genotyping
Clinical Dementia Rating Scale (CDR) | Baseline
  Global cognitive and functional measure
The Activities of Daily Living (ADL) Standardized Scale | Baseline
  Functional measure
Mayo Fluctuations Scale | Baseline
  Behavioral measure
Neuropsychiatric Inventory (NPI) | Baseline
  Behavioral measure
Beck Depression Inventory 2nd ed. | Baseline
  Behavioral measure
The Modified Somatic Perception Questionnaire | Baseline
  Behavioral measure
The Epworth Sleepiness Scale | Baseline
  Sleep measure
Mayo Sleep Questionnaire-Informant | Baseline
  Sleep measure
Functional Outcomes of Sleep Questionnaire-10 | Baseline
  Sleep measure
Part III and IV of the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline
  Gait, Mobility, and Coordination Measure
Berg Balance Scale (BBS) | Baseline
  Gait, Mobility, and Coordination Measure
Florbetapir (F18-AV-45) positron emission tomography (amyloid PET) | Baseline
  Imaging to determine extent of amyloid deposition
Single-photon emission computed tomography (SPECT) with the radioligand [123I]FP-CIT | Baseline
  Functional imaging of the dopamine transporter
Positron emission tomography with 2-(18F) fluoro-2-deoxy-d-glucose (FDG-PET) | Baseline
  Imaging to determine total and regional cerebral glucose metabolism
Brain MRI | Baseline
  Imaging including a resting state functional MRI, diffusion tensor imaging, and anatomic imaging
Polysomnogram | Baseline
  participants will have an overnight standard clinical polysomnogram with added limb leads assessing for presence of sleep apnea, periodic limb movements, and rapid eye movement (REM) sleep characteristics

OTHER OUTCOMES:
Lumbar Puncture to obtain cerebrospinal fluid (CSF) that will be stored for future potential evaluation of biomarkers | Baseline
  Optional outcome measure which will be done to obtain samples of CSF
Post-mortem brain donation to The Ohio State University Neurodegenerative Disease Brain Tissue Repository, for clinicopathological correlations | Post mortem
  Optional outcome measure for patients post-mortem to asses for neuropathologic conditions

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Scharre, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States